CLINICAL TRIAL: NCT06020417
Title: Occurrence of Pedicle Screw Malposition in Spine Arthrodesis Surgeries Performed With O-ARM-guided Navigation at a University Hospital: a Randomized Controlled Trial
Brief Title: Pedicle Screw Malposition in Spine Arthrodesis Surgeries With O-ARM-guided Navigation
Acronym: NoHARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Carlos Eduardo Batista de Lima, MD, PhD, Associate Professor, MD, PhD, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUPiaui_No-HARM
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Spinal Fusion; Spinal Deformity; Spine Injury
Keywords: neuronavigation; spinal deformity; Spine injury
MeSH Terms: conditions — Spinal Injuries | interventions — Arthrodesis

STUDY DESIGN:
Intervention Model Description: Comparison between the use or not of neuronavigation for corrective surgery of spinal deformity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- O-Arm neuronavigator (Active Comparator): The O-ARM imaging system can help surgeons to view the spine in real time and verify the placement of implants such as screws or rods. Primarily, therefore, in image acquisition, during surgery, the O-ARM is activated and generates real-time images of the patient's spine, so that these images are displayed on a screen, allowing the surgeon to visualize the anatomical structures and check that implant placement is proper. Therefore, when analyzing these images, the surgeon can, for example, analyze and verify the placement of the implants and ensure that the arthrodesis is performed correctly, in such a way that, if necessary, the surgeon can make adjustments and then acquire new images for verification.
  Interventions: Device: O-ARM (Medtronic, Inc, Louisville, CO)
- Conventional (Placebo Comparator): The conventional procedure for spinal arthrodesis will involve the intervertebral disc removal step between the vertebrae that will be fused. This is done precisely to create space for the bone graft that will be placed later. Then, there is bone surface preparation, where you prepare the bone surfaces of the vertebrae that will be fused, removing any soft tissue that might interfere with bone fusion. Then, there is bone graft placement, where the surgeon places a bone graft between the vertebrae that will be fused together. This graft can be obtained from another part of the patient's body (such as the pelvis) or from a deceased donor. Then, in the spinal column fixation step, rods, screws and/or plates are used to fix the vertebrae that will be fused.
  Interventions: Procedure: Conventional corrective surgery for arthrodesis

INTERVENTIONS:
Device: O-ARM (Medtronic, Inc, Louisville, CO) — scanner that allows imaging of screws intraoperatively
  Arms: O-Arm neuronavigator
Procedure: Conventional corrective surgery for arthrodesis — Conventional procedure without neuronavigation guide
  Arms: Conventional

SUMMARY:
Background: Throughout the history of spinal deformity there have been continuous advances in the surgical treatment. Although many techniques have been successfully developed despite the anatomy complex, screw placement still remains difficult with a significant risk of misplaced implants. The O-ARM guided Navigation is a scanner that allows imaging of screws intraoperatively and could be a tool to facilitate screw revision and reduce the occurrence of misplaced implants. Methods: This is a prospective and randomized clinical study that will be carried out at the University Hospital of the Federal University of Piaui, which provides exclusive assistance to patients of the Unified Health System (UHS), in northeastern Brazil.

DETAILED DESCRIPTION:
Study design: This is a prospective and randomized clinical study. Local: The study will be carried out at the University Hospital of the Federal University of Piauí (UH-FUPI), which provides exclusive assistance to patients of the Unified Health System (UHS), in the municipality of Teresina (PI), in northeastern Brazil, in the surgical center sector, involving patients undergoing neurosurgical procedures. Data collection will begin after approval by the UH-FUPI research ethics committee. Population and sample: The study population will consist of patients hospitalized for spinal deformities in the wards of the University Hospital of the Federal University of Piauí (UH-FUPI).

Patients aged 18 years or older with surgical indication for spine arthrodesis will be included in the study and will be randomized for corrective neurological or orthopedic spine surgeries performed with O-Arm technology (Intervention Group) and without O-arm (Group control). The surgeries performed electively in the three segments of the spine will be included in this study. Patients who do not sign the informed consent form and those without adequate records in medical records that do not allow the analysis of the data provided for this research will be excluded. Sample size: The sample size of the present study was calculated with the aim of comparing the incidence of misplacement of screws between two approaches, the first using a navigator and the other without. Setting the power of the test at 80% and the confidence level at 95%, the incidence of misplacement of screws known in the literature with the use of a navigator is = 9.8% and without use = 15%. Thus, at least 496 screws would be needed in each arm of the study. Using data from the study by Jin, Liu, Qiu et al. (2017), we noticed that 1145 screws were inserted in 144 patients, generating an average of approximately 8 screws per patient. Thus, at least 62 patients would be needed in each arm. The calculations necessary to determine the sample size were performed by the formula where, is the order percentile of the standard normal distribution, is the order percentile of the standard normal distribution, is the proportion of screw misplacement without using the navigator, is proportion of screw misplacement using the navigator and is the midpoint of the proportions. Data collect: Data will be collected through medical records, which will be completed in the data collection form, after the procedure. The variables analyzed will be: type of surgery performed, technique used, which vertebrae underwent surgical intervention with the implantation of screws, number of screws in each vertebra, presence or not of invasion of the pedicle cortex after analysis with CT, in addition to the description of the affected vertebra , which screws invaded, measurement of invasion, in millimeters, and whether the position was medial or lateral. Statistical analysis: The collected data will be organized in tables and graphs. The program used to carry out the statistical tests will be SPSS Statistics. The method used to jointly analyze the relationship between the studied variables and the presence or absence of expected outcomes will be the Pearson chi-square test method. The admitted confidence interval is 95% and the p-value less than 0.05.

Ethical and legal aspects: All patients included will sign the informed consent form. Data collection will begin after approval of the study by the research ethics committee. All research ethics regulations will be followed according to the resolution of the National Health Council n° 466/12. Risks and benefits: The research risks involve the exposure of personal data and embarrassment to the participants. To work around such problems, patients will be identified by numbering, where only the researchers will have direct access to the patients' records, without photos or any record that could cause the dissemination of personal information. In addition, questions to participants will be asked with caution and empathy, in order to avoid any embarrassment to the patient. If it is demonstrated that the studied neurovagegation system significantly reduces the need for surgical repositioning of the pedicle screws, in addition to the benefit for the sample patient in the intervention group, who will not have to face yet another surgical approach, the FUPI may also be benefited, since the hospital will have, within its list, the option of a neuronavigation technology that brings real results to the hospital's patients.

ELIGIBILITY:
Inclusion Criteria:

* spine deformities (spinal cord trauma, osteoarthritis, intervertebral disc degeneration, degenerative or isthmic spondylolisthesis, intervertebral disc degeneration, spinal stenosis and degenerative scoliosis).

Exclusion Criteria:

* anatomical abnormalities that can not be used the neuronavigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
misplaced implant | 30 days
  medial and/or lateral deviations

SECONDARY OUTCOMES:
recurrent pain | 30 days
  ocurrence of posoperative pain and persistence of symptoms after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Eduardo B Lima, MD, PhD, Principal Investigator — Federal University of Piaui; Denilson G Italiano, Sr., Study Chair — Federal University of Piaui; Mauricio Giraldi, MD, MSc, Study Chair — University Hospital of Federal University of Piaui
Locations (1):
- Carlos Eduardo Batista de Lima, Teresina, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santos ER, Ledonio CG, Castro CA, Truong WH, Sembrano JN. The accuracy of intraoperative O-arm images for the assessment of pedicle screw postion. Spine (Phila Pa 1976). 2012 Jan 15;37(2):E119-25. doi: 10.1097/BRS.0b013e3182257cae. PMID 21673628
- [Background] Perdomo-Pantoja A, Ishida W, Zygourakis C, Holmes C, Iyer RR, Cottrill E, Theodore N, Witham TF, Lo SL. Accuracy of Current Techniques for Placement of Pedicle Screws in the Spine: A Comprehensive Systematic Review and Meta-Analysis of 51,161 Screws. World Neurosurg. 2019 Jun;126:664-678.e3. doi: 10.1016/j.wneu.2019.02.217. Epub 2019 Mar 15. PMID 30880208